CLINICAL TRIAL: NCT00254605
Title: High Resolution Retinal Imaging in Patients With Inherited Retinal Degenerations
Brief Title: Retinal Imaging in Patients With Inherited Retinal Degenerations
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: University of California, Berkeley (Other)
Responsible Party: Sponsor
Other Study IDs: H12225-27221-0+1
Record Dates: First submitted 2005-11-14; First posted 2005-11-16 (Estimated); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Retinitis Pigmentosa
Keywords: imaging; adaptive optics scanning laser ophthalmoscope; optical coherence tomography; electroretinography
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine whether the structure and function of the human retina can be studied with high resolution in patients with inherited retinal degenerations using the Adaptive Optics Scanning Laser Ophthalmoscope (AOSLO).

DETAILED DESCRIPTION:
Retinal degenerations are a group of inherited diseases that result in progressive death of the vision cells, or photoreceptors. Currently there is no treatment or cure for any of these diseases and they ultimately cause blindness in affected patients. We propose to investigate the structure and function of the human retina in patients with inherited retinal degenerations using the Adaptive Optics Scanning Laser Ophthalmoscope (AOSLO). We will correlate the images of retinal structure produced by the AOSLO with Optical Coherence Tomography (OCT) images of the retina. In addition, we will study the vision of individual photoreceptors using the AOSLO to perform a novel technique, microperimetry, in patients with retinal degenerations. We will compare the results of microperimetry with standard measures of vision used in Ophthalmology clinics, including visual acuity, automated perimetry, fundus photography and multifocal electroretinography (mfERG).

The results of this work will provide insight into the mechanism of vision loss among patients with diverse retinal disorders. Specifically, we will study cone structure and function in patients with retinal degenerations with different etiologies: retinitis pigmentosa, a disease usually caused by rod-specific mutations; cone-rod dystrophy, which primarily affects cones rather than rods; and Best's disease, a disease caused by a defect in the retinal pigment epithelium (RPE). In addition, we will study the effect that lipofuscin, a byproduct of photoreceptor metabolism that accumulates in the RPE in diseases such as Stargardt's disease, Best's disease and age-related macular degeneration (AMD), has on cone structure and function, with the goal of understanding how these diseases cause blindness. Better understanding of the mechanisms of vision loss in patients with retinal degeneration should ultimately lead to treatments for these blinding conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must speak and understand English
* Subjects must have pupils that dilate to at least 6 millimeters diameter.
* Subjects must be willing to travel to University of California (UC) Berkeley.
* Subjects are financially responsible for their travel to the San Francisco area if they are not San Francisco residents.

Exclusion Criteria:

* Cataract
* Irregular corneal astigmatism (keratoconus)
* Prior refractive surgery

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with inherited retinal degenerations, including retinitis pigmentosa, choroideremia, x-linked retinoschisis and Usher syndrome. We are also studying a small number of patients with age-related macular degeneration.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2005-11-01; Primary Completion 2028-10 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Cone spacing | 24 months
  The current study will assess cone spacing twice at baseline and every 6 months for 30 months. The primary outcome will be measured at 24 months.

SECONDARY OUTCOMES:
Visual acuity | 24 months
  Visual acuity will be measured every 6 months for 30 months with the primary outcome measure at 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jacque L. Duncan, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- Department of Ophthalmology Retinal Degenerations Clinic, UCSF, San Francisco, California, United States

REFERENCES:
- [Result] Yoon MK, Roorda A, Zhang Y, Nakanishi C, Wong LJ, Zhang Q, Gillum L, Green A, Duncan JL. Adaptive optics scanning laser ophthalmoscopy images in a family with the mitochondrial DNA T8993C mutation. Invest Ophthalmol Vis Sci. 2009 Apr;50(4):1838-47. doi: 10.1167/iovs.08-2029. Epub 2008 Nov 7. PMID 18997096
- [Result] Duncan JL, Zhang Y, Gandhi J, Nakanishi C, Othman M, Branham KE, Swaroop A, Roorda A. High-resolution imaging with adaptive optics in patients with inherited retinal degeneration. Invest Ophthalmol Vis Sci. 2007 Jul;48(7):3283-91. doi: 10.1167/iovs.06-1422. PMID 17591900
- [Result] Roorda A, Zhang Y, Duncan JL. High-resolution in vivo imaging of the RPE mosaic in eyes with retinal disease. Invest Ophthalmol Vis Sci. 2007 May;48(5):2297-303. doi: 10.1167/iovs.06-1450. PMID 17460294
- [Derived] Zayit-Soudry S, Sippl-Swezey N, Porco TC, Lynch SK, Syed R, Ratnam K, Menghini M, Roorda AJ, Duncan JL. Repeatability of Cone Spacing Measures in Eyes With Inherited Retinal Degenerations. Invest Ophthalmol Vis Sci. 2015 Sep 1;56(10):6179-89. doi: 10.1167/iovs.15-17010. PMID 26416092
- [Derived] Wang Q, Tuten WS, Lujan BJ, Holland J, Bernstein PS, Schwartz SD, Duncan JL, Roorda A. Adaptive optics microperimetry and OCT images show preserved function and recovery of cone visibility in macular telangiectasia type 2 retinal lesions. Invest Ophthalmol Vis Sci. 2015 Jan 13;56(2):778-86. doi: 10.1167/iovs.14-15576. PMID 25587056
- [Derived] Menghini M, Lujan BJ, Zayit-Soudry S, Syed R, Porco TC, Bayabo K, Carroll J, Roorda A, Duncan JL. Correlation of outer nuclear layer thickness with cone density values in patients with retinitis pigmentosa and healthy subjects. Invest Ophthalmol Vis Sci. 2014 Dec 16;56(1):372-81. doi: 10.1167/iovs.14-15521. PMID 25515570
- [Derived] Zayit-Soudry S, Duncan JL, Syed R, Menghini M, Roorda AJ. Cone structure imaged with adaptive optics scanning laser ophthalmoscopy in eyes with nonneovascular age-related macular degeneration. Invest Ophthalmol Vis Sci. 2013 Nov 15;54(12):7498-509. doi: 10.1167/iovs.13-12433. PMID 24135755
- [Derived] Ratnam K, Carroll J, Porco TC, Duncan JL, Roorda A. Relationship between foveal cone structure and clinical measures of visual function in patients with inherited retinal degenerations. Invest Ophthalmol Vis Sci. 2013 Aug 28;54(8):5836-47. doi: 10.1167/iovs.13-12557. PMID 23908179
- [Derived] Syed R, Sundquist SM, Ratnam K, Zayit-Soudry S, Zhang Y, Crawford JB, MacDonald IM, Godara P, Rha J, Carroll J, Roorda A, Stepien KE, Duncan JL. High-resolution images of retinal structure in patients with choroideremia. Invest Ophthalmol Vis Sci. 2013 Feb 1;54(2):950-61. doi: 10.1167/iovs.12-10707. PMID 23299470
- [Derived] Ratnam K, Vastinsalo H, Roorda A, Sankila EM, Duncan JL. Cone structure in patients with usher syndrome type III and mutations in the Clarin 1 gene. JAMA Ophthalmol. 2013 Jan;131(1):67-74. doi: 10.1001/2013.jamaophthalmol.2. PMID 22964989
- [Derived] Duncan JL, Ratnam K, Birch DG, Sundquist SM, Lucero AS, Zhang Y, Meltzer M, Smaoui N, Roorda A. Abnormal cone structure in foveal schisis cavities in X-linked retinoschisis from mutations in exon 6 of the RS1 gene. Invest Ophthalmol Vis Sci. 2011 Dec 20;52(13):9614-23. doi: 10.1167/iovs.11-8600. PMID 22110067
- [Derived] Mkrtchyan M, Lujan BJ, Merino D, Thirkill CE, Roorda A, Duncan JL. Outer retinal structure in patients with acute zonal occult outer retinopathy. Am J Ophthalmol. 2012 Apr;153(4):757-68, 768.e1. doi: 10.1016/j.ajo.2011.09.007. Epub 2011 Nov 20. PMID 22105799